CLINICAL TRIAL: NCT01558336
Title: Schistosoma Haematobium Infections Among Schoolchildren in Central Sudan One Year After Treatment With Praziquantel
Brief Title: Schistosoma Haematobium Infections and Praziquantel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Khartoum (Other)
Collaborators: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Principal Investigator, Ishag Adam, Professor, University of Khartoum
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Schistosmiasis
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Schistosomiasis
Keywords: Schistosoma haematobium; schoolchildren; Central Sudan; Praziquantel
MeSH Terms: conditions — Schistosomiasis; Schistosomiasis haematobia | interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Praziguantel (Experimental): tablet single dose
  Interventions: Drug: praziquantel

INTERVENTIONS:
Drug: praziquantel — praziquantel 40 mg/kg oral tablets

SUMMARY:
The purpose of this study is to evaluate the impact of praziquantel for the treatment of Schistosoma haematobium infection among schoolchildren in Al Salamania in Central Sudan.

DETAILED DESCRIPTION:
A longitudinal study will be conducted to evaluate the impact of praziquantel for the treatment of Schistosoma haematobium infection among schoolchildren in Al Salamania in Central Sudan. A cohort of schoolchildren (6-15 years of age) was investigated before and 1 year after treatment with a single dose of praziquantel 40mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* School children

Exclusion Criteria:

* Taking praziquantel

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
cure rate | one year
  The reduction of the prevalence and intensity of S.haematobium infection following a single dose of praziquantel40mg/kg

SECONDARY OUTCOMES:
reduction in the intensity of infection by | one year
  will a single dose of PZQ significantly reduced intensity of infection of S. haematobium infection 1 year after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Al Salamania, Al Salamania, River Nile, Sudan

REFERENCES:
- [Result] Ahmed AM, El Tash LA, Mohamed EY, Adam I. High levels of Schistosoma mansoni infections among schoolchildren in central Sudan one year after treatment with praziquantel. J Helminthol. 2012 Jun;86(2):228-32. doi: 10.1017/S0022149X11000290. Epub 2011 Jun 8. PMID 21729382